CLINICAL TRIAL: NCT05707741
Title: Feasibility of Different Doses of Dexmetomedine to Prevent Post Operative Delirium in Elderly Patients Undergoing Elective Total Knee Replacement Under Spinal Anesthesia
Brief Title: Dexmetomedine for Post Operative Delirium in Elderly Patients Undergoing Elective Total Knee Replacement Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1/2023,ANET2-2
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Delirium
Keywords: Delirium , Dexmetomedine
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: prospective randomized trial
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): normal saline infusion rate 0.4uq/kg /hour
  Interventions: Drug: dexmetomedine infusion
- Group B (Active Comparator): dexmetomedine 0.2 µg/kg/hr
  Interventions: Drug: dexmetomedine infusion
- Group C (Active Comparator): dexmetomedine 0.4 µg/kg/hr
  Interventions: Drug: dexmetomedine infusion

INTERVENTIONS:
Drug: dexmetomedine infusion — 50 ml mixture of saline 49 ml and dexmedetomidine 100 μg,
Drug: Dexmetomedine infusion — 50 ml mixture of saline 48 ml and dexmedetomidine 200 μg

SUMMARY:
Postoperative delirium is a geriatric syndrome occurring after anesthesia and surgery which manifests as acute alterations in mental status, involving changes in cognition, attention, and levels of consciousness that tend to fluctuate The use of dexmedetomidine with the intention to prevent postoperative delirium remains controversial. Where it has shown to be effective in older adult patients undergoing cardiovascular and non-cardiovascular surgeries

DETAILED DESCRIPTION:
On the day of surgery and after arrival to the theatre, all patients will have supplemental oxygen by nasal cannula at 5 L min-1 and will be connected to the standard monitoring non-invasive blood pressure, electrocardiography, and pulse oximetry. crystalloid 10mg/kg will be administered then all patients will receive spinal anaesthesia in the sitting position, under complete aseptic technique. The midline or Para median spinal puncture will be performed. volume of 3 ml of hyperbaric bupivacaine (Marcaine® Spinal Heavy 0.5%, AstraZeneca) will be injected using a 25 G spinal needle . After establishment of spinal anesthesia , A loading dose of dexmetomedine (1 µg/kg) will be administered for 10 min for all the patients then Three types of syringes will be prepared on 50 ml syringes Group A: saline 50 ml, Group B: a 50 ml mixture of saline 49 ml and dexmedetomidine 100 μg, and Group C: a 50 ml mixture of saline 48 ml and dexmedetomidine 200 μg. the patients then they will be randomized into 3 groups

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I- II
* Age from 65to 75 years old,
* Elective total knee arthroplasty under spinal anaesthesia.

Exclusion Criteria:

* Bleeding disorders
* Allergy to any of the drugs used in the study
* Renal insufficiency
* Liver failure-Neurological abnormalities -patients with hearing and visual impairment

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
cognitive functions | 3 days
  Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
Post operative pain | 3days
  VAS (0_10)
Sedation | 3days
  Ramsay sedation score

CONTACTS AND LOCATIONS:
Overall Officials: rabab M habeeb, Dr, Principal Investigator — Menoufia University
Locations (1):
- Menoufia University, Menoufia, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No